CLINICAL TRIAL: NCT03237403
Title: Study of Association Between Clinical Criteria Collected at the SAMU Regulation Centre Call and the Hospital Orientation of Patients With Suspected Sepsis State
Brief Title: Hospital Orientation Since SAMU Regulation Centre Call
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, Romain Jouffroy, Principal Investigator, Hôpital Necker-Enfants Malades
Other Study IDs: 2017-A02335-48
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Sepsis
Keywords: Sepsis; Adults; Pre hospital settings; Triage; Hospital orientation; Outcome
MeSH Terms: conditions — Sepsis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — observational study between clinical criteria collected at SAMU regulation centre call and hospital orientation

SUMMARY:
Specify the association between clinical criteria transmitted by non-medical emergency services to the regulation of the SAMU centre call in patients with suspected sepsis and their hospital orientation: emergency department or intensive care unit

DETAILED DESCRIPTION:
Anonymous, descriptive, longitudinal, resting study searching an association between clinical criteria transmitted by non-medical emergency services to the regulation of the SAMU centre call for patients with suspected sepsis and their subsequent hospital orientation

ELIGIBILITY:
Inclusion Criteria:

* adults (age>18years)
* patients with suspected sepsis state at the regulation SAMU centre call

Exclusion Criteria: minor (age<18years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects calling the SAMU regulation centre call with a clinical suspected sepsis history
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Hospital Admission Service | 1 day
  Emergency department or intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Romain Jouffroy, MD, Principal Investigator — APHP Necker Enfants Malades SAMU 75
Locations (1):
- APHP Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan is planned